CLINICAL TRIAL: NCT06811025
Title: Phase II Clinical Study of Contezolid for the Treatment of Tuberculous Meningitis
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Nie WenJuan, Chief physician, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCP-TB-2024-2-1
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis; Meningitis
Keywords: Tuberculous meningitis; contezolid
MeSH Terms: conditions — Tuberculosis; Meningitis; Tuberculosis, Meningeal | interventions — contezolid; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contezolid (Experimental)
  Interventions: Drug: Contezolid
- linezolid (Active Comparator)
  Interventions: Drug: Linezolid (LZD)

INTERVENTIONS:
Drug: Contezolid — Contezolid 800mg once daily (QD) for 7 days;
  Arms: Contezolid
Drug: Linezolid (LZD) — Linezolid 600mg once daily (QD) for 7 days.
  Arms: linezolid

SUMMARY:
Contezolid is a novel oxazolidinone antibiotic developed by Shanghai Mengke Pharmaceutical Co., Ltd., which successfully went public in 2021. It inhibits bacterial growth by interfering with protein synthesis through its translational inhibitory effect on bacteria. Contezolid has demonstrated promising clinical results in patients with drug-resistant tuberculosis, making it a powerful tool in the fight against drug-resistant tuberculosis.

Currently, there is a lack of pharmacokinetic data on contezolid in patients with central nervous system tuberculosis. Some studies have reported the steady-state concentrations of contezolid in the serum and cerebrospinal fluid (CSF) of tuberculous meningitis patients receiving multidrug therapy, showing that the concentration of contezolid in the CSF exceeds the minimum inhibitory concentration against Mycobacterium tuberculosis, and the unbound fraction has a high penetration rate.

In summary, as a novel anti-tuberculosis drug, contezolid has significant potential value in the treatment of tuberculous meningitis. The implementation of this project will help further explore the application prospects of contezolid in the treatment of tuberculous meningitis and provide a safer and more effective treatment option for clinical use.

DETAILED DESCRIPTION:
Contezolid is a novel oxazolidinone antibiotic developed by Shanghai Mengke Pharmaceutical Co., Ltd., which successfully went public in 2021. It inhibits bacterial growth by interfering with protein synthesis through its translational inhibitory effect on bacteria. Contezolid has demonstrated promising clinical results in patients with drug-resistant tuberculosis, making it a powerful tool in the fight against drug-resistant tuberculosis.

Strong anti-tuberculosis activity: Contezolid exhibits comparable anti-tuberculosis activity to linezolid both in vitro and in vivo, and even superior intracellular bactericidal activity against Mycobacterium tuberculosis.

High safety: Contezolid significantly reduces the risks of bone marrow suppression toxicity, neurotoxicity, and lactic acidosis compared to linezolid, bringing new hope to patients who cannot continue traditional therapy due to adverse drug reactions.

Broad application prospects: With the further accumulation of clinical data and in-depth research, the application prospects of contezolid in anti-tuberculosis treatment will undoubtedly be broader. Especially for patients who experience severe adverse reactions and cannot continue using linezolid, contezolid provides a new treatment option.

Currently, there is a lack of pharmacokinetic data on contezolid in patients with central nervous system tuberculosis. Some studies have reported the steady-state concentrations of contezolid in the serum and cerebrospinal fluid (CSF) of tuberculous meningitis patients receiving multidrug therapy, showing that the concentration of contezolid in the CSF exceeds the minimum inhibitory concentration against Mycobacterium tuberculosis, and the unbound fraction has a high penetration rate.

In summary, as a novel anti-tuberculosis drug, contezolid has significant potential value in the treatment of tuberculous meningitis. The implementation of this project will help further explore the application prospects of contezolid in the treatment of tuberculous meningitis and provide a safer and more effective treatment option for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* (1) Inpatients who have been diagnosed with or clinically diagnosed with tuberculous meningitis within the past 3 months prior to screening; (2) Voluntarily participate in this study and sign the informed consent form; (3) Male and female participants must use effective contraception during the study and for 1 month after the study ends.

Exclusion Criteria:

* (1) Patients who have been on long-term corticosteroid therapy or taking immunosuppressants within 90 days prior to screening; (2) Pregnant women, patients in the puerperium, and lactating women; (3) Patients with a history of allergy or known hypersensitivity to contezolid or linezolid, or a history of severe adverse reactions; (4) Patients with evidence of resistance to contezolid or linezolid; (5) Patients deemed unsuitable for participation in this study by the investigator's assessment; (6) Patients whom the investigator believes participation in this study would harm their health, or who are deemed unable to comply with the scheduled visits and assessments as outlined in the protocol, and therefore unsuitable for participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
After 7 days of oral treatment with contezolid/linezolid, the patients underwent lumbar puncture to obtain cerebrospinal fluid (CSF) samples, and concentration tests were conducted on both blood and CSF samples. | 7 days
  After 7 days of oral treatment with contezolid/linezolid, the patients underwent lumbar puncture to obtain cerebrospinal fluid (CSF) samples, and concentration tests were conducted on both blood and CSF samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chest hospital affiliated to Capital medical university, Beijing Tuberculosis & Thoracic Tumor Research Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In our institution, it is not allowed to post hospital information and patient information on websites for public disclosure.